CLINICAL TRIAL: NCT04626310
Title: Mapping Treatment Components to Targets in Dialectical Behavior Therapy
Brief Title: Mapping Aspects of Psychotherapy in Dialectical Behavior Therapy
Acronym: MAP-DBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Toledo (Other)
Responsible Party: Principal Investigator, Katherine Dixon-Gordon, Associate Professor, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1710 1R21MH119530-01A1; R21MH119530-01A1 (NIH)
Record Dates: First submitted 2020-11-01; First posted 2020-11-12 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Borderline Personality Disorder
Keywords: Dialectical behavior therapy; Emotions; Behavior and Behavior mechanisms; Randomized Controlled Trials
MeSH Terms: conditions — Borderline Personality Disorder; Behavior | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dialectical behavior therapy - emotion regulation skills training (Experimental): Dialectical behavior therapy - emotion regulation skills training
  Interventions: Behavioral: Dialectical behavior therapy - emotion regulation skills training
- Dialectical behavior therapy - interpersonal effectiveness skills training (Experimental): Dialectical behavior therapy - interpersonal effectiveness skills training
  Interventions: Behavioral: Dialectical behavior therapy - interpersonal effectiveness skills training
- Non-skills-oriented interpersonal psychotherapy group (Active Comparator): Non-skills-oriented interpersonal psychotherapy group
  Interventions: Behavioral: Interpersonal psychotherapy

INTERVENTIONS:
Behavioral: Dialectical behavior therapy - emotion regulation skills training — Arm 1. Dialectical behavior therapy - emotion regulation skills training follows the emotion regulation skills DBT Skills Training Manual Second Edition and the DBT Skills Training Handouts and Worksheets Second Edition. This group involves 6 weekly sessions.
  Arm 2. Dialectical behavior therapy - interpersonal effectiveness skills training follows the interpersonal effectiveness skills DBT Skills Training Manual Second Edition and the DBT Skills Training Handouts and Worksheets Second Edition. This group involves 6 weekly sessions.
  Arms: Dialectical behavior therapy - emotion regulation skills training
Behavioral: Dialectical behavior therapy - interpersonal effectiveness skills training — Arm 2. Dialectical behavior therapy - interpersonal effectiveness skills training follows the interpersonal effectiveness skills DBT Skills Training Manual Second Edition and the DBT Skills Training Handouts and Worksheets Second Edition. This group involves 6 weekly sessions.
  Arms: Dialectical behavior therapy - interpersonal effectiveness skills training
Behavioral: Interpersonal psychotherapy — Arm 3. Non-skills-oriented interpersonal psychotherapy group follows evidence-based principles on common factors in a group therapy context. This group involves 6 weekly sessions.
  Arms: Non-skills-oriented interpersonal psychotherapy group

SUMMARY:
Although dialectical behavior therapy (DBT) skills training is effective in the treatment of borderline personality disorder, it contains four skills modules and there is little research to guide their modular application. This study compares the unique effects of two distinct DBT skills training modules, relative to a non-DBT therapy group for adults with borderline personality disorder. Using innovative laboratory-based assessment methods, the proposed study will examine the effects of these conditions on emotional responding and interpersonal functioning, as well as clinical outcomes.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a severe mental health condition with high morbidity and mortality. Although dialectical behavior therapy (DBT) is an efficacious treatment for BPD, it is resource-intensive and lengthy in its full form, involving one year of weekly individual therapy and group skills training in mindfulness, emotion regulation, interpersonal effectiveness, and distress tolerance. As a result, few patients have access to the full treatment. A better understanding of how the distinct components of DBT affect different sets of symptoms could help to streamline this treatment and personalize its use with specific patients.

Improvements in both interpersonal and emotional functioning are theorized to underlie improvements in BPD. Thus, emotion regulation and interpersonal effectiveness skills training may be particularly important components of DBT. Therefore, this study examines the unique effects of two distinct DBT skills training modules.

Participants are adults with BPD and recent, recurrent self-injurious behaviors (planned N = 81) who are randomly assigned to six weeks of DBT emotion regulation skills training (DBT-ER), DBT interpersonal effectiveness skills training (DBT-IE), or a non-skills control group. Using innovative laboratory-based multimethod assessments, this study examines the effects of these conditions on emotional responding and interpersonal functioning, as well as BPD related outcomes. Aim 1 examines the unique effects of DBT-ER and DBT-IE on their respective emotion-related (subjective and biological emotional reactivity, behavioral emotion regulation, skills use) and interpersonal (subjective and behavioral) targets, compared to the non-DBT treatment. Aim 2 examines whether improved emotional functioning predicts reductions in BPD symptoms and self-injury. Aim 3 examines whether baseline emotion dysregulation interacts with treatment condition to predict treatment response.

The proposed research is innovative in its experimental examination of the effects of DBT components on specific targets in BPD. Given the high societal costs of BPD, this work has important public health significance. Findings will inform larger studies evaluating the potential modular use of DBT components to result in briefer and more efficient individualized treatments for patients.

ELIGIBILITY:
Inclusion Criteria:

1. exhibit 4+ BPD symptoms,
2. have a history of recent (i.e., past-year) and recurrent (> 1 instance) of self-injury,
3. commit to participate in one of our 6-week experimental groups,
4. have an individual health provider who can manage imminent issues,
5. be between 18-60 years old,

Exclusion Criteria:

1. not fluent in English,
2. have impaired (uncorrected) vision or hearing that would impair ability to understand study stimuli,
3. a current manic, psychotic, or active physiological dependence on substances (to limit interference in the lab),
4. low cognitive functioning (IQ ≤ 70.4 (TOPF; Pearson Assessments, 2009),
5. past DBT treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Dixon-Gordon, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- Psychological Services Center, University of Massachusetts Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via NDA.
Time Frame: Data are expected to be cleaned scored and uploaded by Jan 2024
Access Criteria: Data will be available through NDA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: N=115 recruited from the area around western MA assessed for eligibility but only 84 enrolled in study. .
Pre-assignment Details: Due to group design, participants waited for next group date to begin treatment
Groups:
- Dialectical Behavior Therapy - Emotion Regulation Skills Training: Dialectical behavior therapy - emotion regulation skills training
  Dialectical behavior therapy - emotion regulation skills training: Arm 1. Dialectical behavior therapy - emotion regulation skills training follows the emotion regulation skills DBT Skills Training Manual Second Edition and the DBT Skills Training Handouts and Worksheets Second Edition. This group involves 6 weekly sessions.
  Arm 2. Dialectical behavior therapy - interpersonal effectiveness skills training follows the interpersonal effectiveness skills DBT Skills Training Manual Second Edition and the DBT Skills Training Handouts and Worksheets Second Edition. This group involves 6 weekly sessions.
Period: Overall Study
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Started | 27 | 28 | 29
Completed | 20 | 23 | 21
Not Completed | 7 | 5 | 8
Not completed — 4-miss from treatment | 6 | 5 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group | Total
Number analyzed (Participants) | 27 | 28 | 29 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 28 | 29 | 84
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.41 (11.71) | 25.75 (9.95) | 24.72 (7.21) | 25.61 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 25 | 75
  Male | 3 | 2 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 1 | 8
  Not Hispanic or Latino | 22 | 26 | 28 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 5 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 15 | 20 | 22 | 57
  More than one race | 4 | 2 | 0 | 6
  Unknown or Not Reported | 3 | 1 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 29 | 84
DERS total [Mean (Standard Deviation); unit: units on a scale] — Population: Means are provided separately for DBT-ER (n = 27), DBT-IE (n = 28), and interpersonal psychotherapy (n = 29)
  units on a scale | 118.525 (23.707) | 116.539 (21.399) | 120.915 (23.707) | 118.688 (21.363)

OUTCOME MEASURES:

1. Primary Outcome: Change in Emotional Functioning - Linear
Description: Assessed with the Difficulties in Emotion Regulation Scale (DERS), which has total scores that range from 36-180, with higher scores indicating more difficulties. Outcomes are reported as slopes (scores over weeks, centered around the start of treatment, with standard errors) per condition, extracted from mixed effects/multilevel models. This measure is listed separately to permit presentation of two units of measure (that are in the same model) - the Linear unit of measure (DERS scores/week), and the Quadratic unit of measure (DERS scores/week^2). This measure reflects the Linear measure.
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7, follow-up week 13-14
Population: ITT sample (see study description)
Measure: Mean (Standard Error); unit: DERS scores/wk
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 27 | 28 | 29
DERS scores/wk | -.917 (.31) | -1.25 (.32) | -1.01 (.26)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Comparisons of Linear Slopes (DBT-ER vs. IP) in latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) with quadratic effects; Test type: Superiority; p = .8, Mixed Models Analysis; Linear slope difference DBT-ER-IP = .096, Standard Error of Mean .08
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Comparisons of Linear Slopes (DBT-IE vs. IP) in latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) with quadratic effects; Test type: Superiority; p = .544, Mixed Models Analysis; Linear Slope difference DBT-IE-IP = -0.234, Standard Error of Mean .385
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Comparisons of Linear Slopes (DBT-ER vs. DBT-IE) in latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) with quadratic effects; Test type: Superiority; p = .442, Mixed Models Analysis; Linear Slope difference DBT-ER-DBT-IE = .329, Standard Error of Mean .429

2. Primary Outcome: Change in Borderline Personality Disorder Features - Linear
Description: Assessed with the abbreviated Borderline Symptom List (BSL23), which has mean scores that range from 0-4, with higher scores indicating more symptoms. Outcomes are reported as slopes (scores rescaled *100 over weeks, centered around the start of treatment, with standard errors) per condition, extracted from mixed effects/multilevel models. This measure is listed separately to permit presentation of two units of measure (that are in the same model) - the Linear unit of measure (BSL scores/week), and the Quadratic unit of measure (BSL scores/week^2). This measure reflects the Linear measure.
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7, follow-up week 13-14
Population: missing 1 data point for DBT-ER group
Measure: Mean (Standard Error); unit: BSL scores/wk
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 26 | 28 | 29
BSL scores/wk | -1.716 (.808) | -3.567 (.746) | -3.667 (.833)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .09, Mixed Models Analysis; Linear slope difference DBT-ER-IP = 1.951, Standard Error of Mean 1.15
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = .93, Mixed Models Analysis; Linear slope difference DBT-IE-IP = .100, Standard Error of Mean 1.228
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = .93, Mixed Models Analysis; Linear slope difference DBT-ER-DBT-IE = 1.851, Standard Error of Mean 1.103
Statistical Analysis 4: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Comparisons of Quadratic Slopes (DBT-ER vs. IP) in latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) with quadratic effects; Test type: Superiority; p = .93, Mixed Models Analysis; Quad slope difference DBT-ER-IP = -.028, Standard Error of Mean .15
Statistical Analysis 5: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Comparisons of Quadratic Slopes (DBT-IE vs. IP) in latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) with quadratic effects; Test type: Superiority; p = .836, Mixed Models Analysis; Quad slope difference DBT-IE-IP = -.029, Standard Error of Mean .145
Statistical Analysis 6: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = .994, Mixed Models Analysis; Quad slope difference DBT-ER-DBT-IE = .001, Standard Error of Mean .145

3. Secondary Outcome: Change in Self-reported Emotional Reactivity
Description: Assessed with self-reported emotions on the PANAS negative affect (NA) scale (mean scores on a scale of 1-5) in response to emotional scripts (Neg: neutral (Neu), negative (Neg)) by emotion regulation condition (Reg: emotional maintain instructions, and negative with decrease instructions) presented in the lab. Outcomes are reported as slopes differences in PANAS NA scores between neutral and negative-maintain over weeks (centered around the start of treatment, with standard errors) per condition, extracted from mixed effects/multilevel models.
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7
Measure: Mean (Standard Error); unit: Condition diff (Neg-Neu) in NA scores/wk
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 27 | 28 | 29
Condition diff (Neg-Neu) in NA scores/wk | -.07 (.06) | -.09 (.06) | -.12 (.06)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. The slopes of the difference between neutral and negative-maintain were regressed on time (weeks, centered around the start of treatment) and calculated per condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to IP; Test type: Superiority; p = .475, Mixed Models Analysis; Linear slope difference DBT-ER-IP = .059, Standard Error of Mean .083
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. The slopes of the difference between neutral and negative-maintain were regressed on time (weeks, centered around the start of treatment) and calculated per condition. Models tested whether these slopes differed by condition. This test compared DBT-IE to IP; Test type: Superiority; p = .654, Mixed Models Analysis; Linear slope difference DBT-IE-IP = .037, Standard Error of Mean .082
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. The slopes of the difference between neutral and negative-maintain were regressed on time (weeks, centered around the start of treatment) and calculated per condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to DBT-IE; Test type: Superiority; p = .791, Mixed Models Analysis; Linear slope difference DBT-ER-DBT-IE = .022, Standard Error of Mean .085

4. Secondary Outcome: Change in Self-reported Emotional Regulation
Description: Assessed with self-reported emotions on the PANAS negative affect (NA) scale (mean scores on a scale of 1-5) in response to emotional scripts (neutral (Neu), negative (Neg)) by emotion regulation condition (Reg: with emotional maintain (Main) instructions, and negative with decrease (Dec) instructions) presented in the lab. Outcomes are reported as slopes differences in PANAS NA scores between Reg conditions in response to negative stimuli (negative-decrease and negative-maintain) over weeks (centered around the start of treatment, with standard errors) per condition, extracted from mixed effects/ multilevel models.
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7
Measure: Mean (Standard Error); unit: Condition diff (Reg) in NA score/wk
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 27 | 28 | 29
Condition diff (Reg) in NA score/wk | -.18 (.07) | -.01 (.07) | .15 (.07)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. We examined the effect of Negative Decrease vs. Negative Maintain over time per condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to IP; Test type: Superiority; p = .001, Mixed Models Analysis; Linear slope difference DBT-ER-IP = -.332, Standard Error of Mean .095
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. We examined the effect of Negative Decrease vs. Negative Maintain over time per condition. Models tested whether these slopes differed by condition. This test compared DBT-IE to IP; Test type: Superiority; p = .078, Mixed Models Analysis; Linear slope difference DBT-IE-IP = -.165, Standard Error of Mean .094
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. We examined the effect of Negative Decrease vs. Negative Maintain over time per condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to DBT-IE; Test type: Superiority; p = .080, Mixed Models Analysis; Linear slope difference DBT-ER-DBT-IE = -.167, Standard Error of Mean .095

5. Secondary Outcome: Change in Affect-modulated Startle
Description: Assessed with eyeblink startle amplitude (mV) in response to emotional cues presented in the lab (of note, per protocol, we examined eyeblink in response to negative and neutral image stimuli across initial [novel] and repeated presentations) which were presented along with sound bursts to elicit startle. This outcome was transformed and then rescaled (*100, = mVtr). Outcomes are reported as slopes per condition over weeks (centered around the start of treatment, with standard errors) per condition, extracted from mixed effects/multilevel models with image valence (Neg: negative vs. neutral) and type (Novel: novel vs. repeated) within-person condition effects.
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7
Population: Some participants were missing data due to nonattendance at lab sessions
Measure: Mean (Standard Error); unit: Condition diff (NegXNovel) in Mn mVtr/Wk
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 25 | 25 | 25
Condition diff (NegXNovel) in Mn mVtr/Wk | .015 (.041) | .043 (.040) | -.076 (.044)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. The Negative x Novel x time (weeks, centered around the start of treatment) slopes were calculated per condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to IP; Test type: Superiority; p = .13, Mixed Models Analysis; Linear Slope Diff DBT-ER-IP = .091, Standard Error of Mean .06
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. The Negative x Novel x time (weeks, centered around the start of treatment) slopes were calculated per condition. Models tested whether these slopes differed by condition. This test compared DBT-IE to IP; Test type: Superiority; p = .046, Mixed Models Analysis; Linear slope difference DBT-IE-IP = .12, Standard Error of Mean .06
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. The Negative x Novel x time (weeks, centered around the start of treatment) slopes were calculated per condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to DBT-IE; Test type: Superiority; p = .617, Mixed Models Analysis; Linear slope difference DBT-ER-DBT-IE = -.028, Standard Error of Mean .057

6. Secondary Outcome: Change in Emotional Habituation
Description: Assessed with skin conductance (SC; microsiemens, μS) in response to emotional cues presented in the lab (of note, per protocol, we examined DV in response to negative and neutral image stimuli [Neg] across initial [Novel] and repeated presentations) which were presented along with sound bursts to elicit startle. Data were transformed to address skew (μStr). Outcomes are reported as novel x negative slopes (SLP) over weeks (centered around the start of treatment, with standard errors) per condition, extracted from mixed effects / multilevel models.
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7
Population: Missing data due to nonattendance at lab visits
Measure: Mean (Standard Error); unit: Condition diff (NegxNovel) in Mn μStr/wk
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 25 | 25 | 25
Condition diff (NegxNovel) in Mn μStr/wk | -.156 (.07) | .023 (.069) | .134 (.076)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of change in this interaction effect were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to IP; Test type: Superiority; p = .005, Mixed Models Analysis; Linear slope difference DBT-ER-IP = -.29, Standard Error of Mean .103
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of change in this interaction effect were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-IE to IP; Test type: Superiority; p = .281, Mixed Models Analysis; Linear slope difference DBT-IE-IP = -.111, Standard Error of Mean .103
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of change in this interaction effect were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to DBT-IE; Test type: Superiority; p = .066, Mixed Models Analysis; Linear slope difference DBT-ER-DBT-IE = -.18, Standard Error of Mean .098

7. Secondary Outcome: Change in Physiological Emotional Reactivity
Description: Assessed with skin conductance (SC; microsiemens, μS) in response to emotional scripts (Neg: neutral, negative) by emotion regulation (Reg: emotional maintain instructions, and negative with decrease instructions) presented in the lab. Data were transformed to address skew (μStr). Outcomes are reported as slopes of Negative (Neg) condition effects on SC over weeks (centered around the start of treatment, with standard errors) per condition, extracted from mixed effects / multilevel models.
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7
Measure: Mean (Standard Error); unit: Condition diff (Neg) in Mean μS/week
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 27 | 28 | 29
Condition diff (Neg) in Mean μS/week | 1.46 (.48) | -.71 (.4) | .41 (.39)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of the effect of negative maintain vs. neutral images on weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to IP; Test type: Superiority; p = .108, Mixed Models Analysis; Linear slope difference DBT-ER-IP = 1.049, Standard Error of Mean .653
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of the effect of negative maintain vs. neutral images on weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-IE to IP; Test type: Superiority; p = .014, Mixed Models Analysis; Linear slope difference DBT-IE-IP = -1.21, Standard Error of Mean .454
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of the effect of negative maintain vs. neutral images on weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to DBT-IE; Test type: Superiority; p = .001, Mixed Models Analysis; Linear slope difference DBT-ER-DBT-IE = 2.17, Standard Error of Mean .631

8. Secondary Outcome: Change in Deliberate Physiological Emotional Regulation
Description: Assessed with high frequency heart rate variability (HRV, ms2/hz) in response to emotional scripts (Negative: negative vs. neutral) with emotion regulation instructions (Reg: Maintain vs. Decrease in the Negative condition) presented in the lab. Data were transformed to address skew (ms2/hztr). Outcomes are reported as slopes of the effect of the Reg condition on HRV over weeks (centered around the start of treatment, with standard errors) per condition, extracted from mixed effects /multilevel models.
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7
Measure: Mean (Standard Error); unit: Condition diff (Reg) on Mn ms2/hztr/week
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 27 | 28 | 29
Condition diff (Reg) on Mn ms2/hztr/week | .08 (.1) | .10 (.10) | .10 (.09)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of the effect of negative maintain vs. negative decrease on weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to IP; Test type: Other; p = .211, Mixed Models Analysis; Linear Slope difference DBT-ER-IP = .17, Standard Error of Mean .136
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of the effect of negative maintain vs. negative decrease on weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-IE to IP; Test type: Superiority; p = .148, Mixed Models Analysis; Linear Slope difference DBT-IE-IP = -.195, Standard Error of Mean .135
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of the effect of negative maintain vs. negative decrease on weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to DBT-IE; Test type: Superiority; p = .857, Mixed Models Analysis; Linear Slope difference DBT-ER-DBT-IE = -.025, Standard Error of Mean .137

9. Other Pre Specified Outcome: Change in Coping Strategies - Linear
Description: Assessed with the DBT-Ways of Coping Checklist (DBT-WCCL, transformed = DBTWCCLtr), which yields scales of skills use (DSS, rescaled *100), general dysfunctional coping (DC1, rescaled *10), and blaming others (DC2, *10), with scores of 0-3, higher reflects greater use. Outcomes are reported as slopes (with SE) centered around treatment start per condition, extracted from mixed effects/multilevel models (separately per scale score).This measure is listed separately to permit presentation of two units of measure (that are in the same model) for the DC1 scale, which was fit best with a quadratic model, whereas the remaining scales only required a Linear model. This measure reflects the Linear measures (DBTWCCL/week) for all scales.
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7, follow-up week 13-14
Measure: Mean (Standard Error); unit: DBTWCCLtr scores/week
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 27 | 28 | 29
DBTWCCLtr scores/week
  DSS - Linear ONLY - rescaled *100 | .23 (.559) | .546 (.523) | .544 (.562)
  DC1 - Linear - rescaled *10 | -.17 (.08) | -.31 (.07) | -.26 (.07)
  DC2 - Linear ONLY- rescaled *10 | -.174 (.079) | -.230 (.074) | -.219 (.080)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DSS over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to IP; Test type: Superiority; p = .693, Mixed Models Analysis; Linear Slope Difference in DSS DBT-ER-IP = -.313, Standard Error of Mean .794
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DSS over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-IE to IP; Test type: Superiority; p = .998, Mixed Models Analysis; Linear Slope Difference in DSS DBT-IE-IP = .002, Standard Error of Mean .767
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DSS over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to DBT-IE; Test type: Superiority; p = .680, Mixed Models Analysis; Linear Slope Diff in DSS DBT-ER-DBT-IE = -.315, Standard Error of Mean .765
Statistical Analysis 4: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DC1 over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-ER to IP; Test type: Superiority; p = .333, Mixed Models Analysis; Linear Slope Difference in DC1 DBT-ER-IP = .098, Standard Error of Mean .101
Statistical Analysis 5: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DC1 over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-IE to IP; Test type: Superiority; p = .632, Mixed Models Analysis; Linear Slope Diff in DC1 DBT-IE-IP = -.046, Standard Error of Mean .097
Statistical Analysis 6: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DC1 over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared DBT-IE to DBT-ER; Test type: Superiority; p = .178, Mixed Models Analysis; Linear Slope Diff in DC1 DBT-ER-DBT-IE = .144, Standard Error of Mean .107
Statistical Analysis 7: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DC2 over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared the slope differences DBT-ER to IP; Test type: Superiority; p = .689, Mixed Models Analysis; Linear Slope Diff in DC2 DBT-ER-IP = .045, Standard Error of Mean .112
Statistical Analysis 8: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DC2 over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared the slope differences DBT-IE to IP; Test type: Superiority; p = .917, Mixed Models Analysis; Linear Slope Diff in DC2 DBT-IE-IP = -.011, Standard Error of Mean .109
Statistical Analysis 9: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DC2 over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared the slope differences DBT-ER to DBT-IE; Test type: Superiority; p = .603, Mixed Models Analysis; Linear Slope Diff in DC2 DBT-ER-DBT-IE = .056, Standard Error of Mean .108

10. Primary Outcome: Change in Emotional Functioning - Quad
Description: Assessed with the Difficulties in Emotion Regulation Scale (DERS), which has total scores that range from 36-180, with higher scores indicating more difficulties. Outcomes are reported as slopes (scores over weeks, centered around the start of treatment, with standard errors) per condition, extracted from mixed effects/multilevel models. This measure is listed separately to permit presentation of two units of measure (that are in the same model) - the Linear unit of measure (DERS scores/week), and the Quadratic unit of measure (DERS scores/week^2). This measure reflects the Quadratic measure.
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7, follow-up week 13-14
Population: ITT sample (see study description)
Measure: Mean (Standard Error); unit: DERS scores/wk^2
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 27 | 28 | 29
DERS scores/wk^2 | -.06 (.04) | -.04 (.04) | -.07 (.03)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = .762, Mixed Models Analysis; Other[Quad Slope difference DBT-ER-IP] = .013, Standard Error of Mean .044
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = .478, Mixed Models Analysis; Quad Slope difference DBT-IE-IP = .034, Standard Error of Mean .047
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Comparisons of Quadratic Slopes (DBT-ER vs. DBT-IE) in latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) with quadratic effects; Test type: Superiority; p = .705, Mixed Models Analysis; Quad Slope difference DBT-ER-DBT-IE = -.089, Standard Error of Mean .054

11. Primary Outcome: Change in Borderline Personality Disorder Features - Quad
Description: Assessed with the abbreviated Borderline Symptom List (BSL23), which has mean scores that range from 0-4, with higher scores indicating more symptoms. Outcomes are reported as slopes (scores rescaled *100 over weeks, centered around the start of treatment, with standard errors) per condition, extracted from mixed effects/multilevel models. This measure is listed separately to permit presentation of two units of measure (that are in the same model) - the Linear unit of measure (BSL scores/week), and the Quadratic unit of measure (BSL scores/week^2). This measure reflects the Quadratic measure.
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7, follow-up week 13-14
Population: missing 1 data point for DBT-ER group from ITT sample
Measure: Mean (Standard Error); unit: BSL scores/wk^2
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 26 | 28 | 29
BSL scores/wk^2 | -.162 (.108) | -.163 (.095) | -.135 (.100)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = .93, Mixed Models Analysis; Quad slope difference DBT-ER-IP = -.028, Standard Error of Mean .15
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = .836, Mixed Models Analysis; Quad slope difference DBT-IE-IP = -.029, Standard Error of Mean .145
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = .994, Mixed Models Analysis; Quad slope difference DBT-ER-DBT-IE = .001, Standard Error of Mean .145

12. Other Pre Specified Outcome: Change in Coping Strategies - Quad
Description: Assessed with the DBT-Ways of Coping Checklist (DBT-WCCL, transformed = DBTWCCLtr), which yields scales of skills use (DSS, rescaled *100), general dysfunctional coping (DC1, rescaled *10), and blaming others (DC2, *10), with scores of 0-3, higher reflects greater use. Outcomes are reported as slopes (SE) centered around treatment start per condition, extracted from mixed effects/multilevel models (separately per scale score).This measure is listed separately to permit presentation of two units of measure (that are in the same model) for the DC1 scale, which was fit best with a quadratic model, whereas the remaining scales only required a Linear model. This measure reflects the Quadratic measure (DBTWCCL/week^2).
Time Frame: Pre-treatment, mid-treatment week 3-4, post-treatment week 6-7, follow-up week 13-14
Population: ITT sample
Measure: Mean (Standard Error); unit: DBTWCCLtr DC1 scores/week^2
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
Number analyzed (Participants) | 27 | 28 | 29
DBTWCCLtr DC1 scores/week^2 | -002 (.011) | -.012 (.007) | -.015 (.007)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DC1 over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared the quadratic effects differed DBT-ER to IP; Test type: Superiority; p = .313, Mixed Models Analysis; Quad slope diff in DC1 DBT-ER-IP = .013, Standard Error of Mean .013
Statistical Analysis 2: Comparison: Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training vs Non-skills-oriented Interpersonal Psychotherapy Group; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DC1 over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared the quadratic effects differed DBT-IE to IP; Test type: Superiority; p = .747, Mixed Models Analysis; Quad Slope in DC1 DBT-IE-IP = .003, Standard Error of Mean .01
Statistical Analysis 3: Comparison: Dialectical Behavior Therapy - Emotion Regulation Skills Training vs Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training; Latent growth curve models (in multilevel/mixed effects framework, Mplus v8.1) were estimated with maximum likelihood. Simple slopes of DC1 over weeks were calculated for each condition. Models tested whether these slopes differed by condition. This test compared the quadratic effects differed DBT-ER to DBT-IE; Test type: Superiority; p = .444, Mixed Models Analysis; Quad slope diff in DC1 DBT-ER-DBT-IE = .009, Standard Error of Mean .012

ADVERSE EVENTS:
Time Frame: Baseline to 13-14 wk timepoint
Arm/Group | Dialectical Behavior Therapy - Emotion Regulation Skills Training | Dialectical Behavior Therapy - Interpersonal Effectiveness Skills Training | Non-skills-oriented Interpersonal Psychotherapy Group
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 0/29

LIMITATIONS AND CAVEATS:
Please note that initial results have not yet been peer-reviewed. As a pilot study conducted during COVID, this study was pivoted to offer telehealth during a time of social distancing. This likely increased amount of missing data for in-person assessed visits. Relatively low power for mixed effects models suggest alternative approaches to data analysis may need to be considered, but initial trial results are presented as originally proposed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT04626310/Prot_SAP_000.pdf